CLINICAL TRIAL: NCT06039826
Title: A Phase 1 Study to Investigate the Effect of LY3437943 on the Pharmacokinetics of the Combined Oral Contraceptive Ethinyl Estradiol and Drospirenone in Female Participants
Brief Title: A Study of LY3437943 in Postmenopausal Female Participants Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18533; J1I-MC-GZBV (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-09-11; First posted 2023-09-15 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Overweight
Keywords: Pharmacokinetics; Obesity; Oral Contraceptive
MeSH Terms: conditions — Overweight; Obesity | interventions — retatrutide; Ethinyl Estradiol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3437943 + Combined Oral Contraceptive (COC) (Experimental): The COC ethinyl estradiol and drospirenone administered orally in combination with LY3437943 administered subcutaneously (SC).
  Interventions: Drug: LY3437943; Drug: Ethinyl Estradiol; Drug: Drospirenone

INTERVENTIONS:
Drug: LY3437943 — Administered SC.
Drug: Ethinyl Estradiol — Administered orally
Drug: Drospirenone — Administered orally

SUMMARY:
The main purpose of this study is to determine the effect of LY3437943 when administered subcutaneously on the levels of combined oral contraceptive (COC) ethinyl estradiol and drospirenone in the blood stream in postmenopausal female participants who are overweight or obese. The safety and tolerability of LY3437943 when administered with COC will also be evaluated. This study will last up to approximately 29 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female participants
* Body mass index (BMI) within the range 27.0 to 40.0 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have an unstable disease or a disease constituting a risk when taking the study intervention.
* Have significant renal insufficiency
* Have an important gastro-esophageal reflux disease, pyloric stenosis, gastroparesis or a history of gastric bypass surgery.
* Have a history or presence of chronic or idiopathic acute pancreatitis.
* Have a history of severe clinically significant multiple or severe drug allergies.
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
* Have had any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin or in situ carcinoma of the cervix that have been resected with no evidence of metastatic disease for 3 years
* Have any form of diabetes mellitus other than type 2
* Have type 2 diabetes with HbA1c greater than or equal to 10% at screening
* Have received an oral or transdermal patch hormone replacement therapy (HRT) within the last 1 month prior to screening or depot injectable HRT within the last 6 months
* Have received any investigational drug within the last month or 5 half-lives of this drug, whichever is longer, prior to screening. If the half-life of the previous investigational drug is unknown, the washout period should be at least 3 months before screening
* Show evidence of HIV infection or positive HIV antibodies
* Have evidence of, or test positive for, anti-hepatitis C virus antibody unless a confirmatory test for hepatitis C virus RNA is negative
* Test positive for hepatitis B surface antigen. In case a hepatitis B virus DNA test was also performed recently and is positive, the participant should be excluded independently of the hepatitis B surface antigen test result. The hepatitis B core antibody test is not used to assess eligibility
* Have acute or chronic hepatitis, or signs and symptoms of any other liver disease, or with significant abnormalities in laboratory liver tests
* Have a fasting triglyceride level greater than 500 mg/dL at screening
* Used any nicotine product including tobacco or nicotine replacement products within 1 month prior to screening or a positive cotinine test at screening. Are unable or unwilling to refrain from using such products during the study
* Have donated at least 450 mL of blood within 8 weeks before screening or intend to donate blood during the study

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time zero to 24 Hours Postdose (AUC0-24) of Ethinyl Estradiol | Predose on Day 1 up to 144 days postdose
  PK: AUC0-24 of Ethinyl Estradiol
PK: Maximum Observed Concentration (Cmax) of Ethinyl Estradiol | Predose on Day 1 up to 144 days postdose
  PK: Cmax of Ethinyl Estradiol
PK: Time of Maximum Observed Concentration (Tmax) of Ethinyl Estradiol | Predose on Day 1 up to 144 days postdose
  PK: Tmax of Ethinyl Estradiol
PK: Area Under the Concentration Versus Time Curve from Time zero to 24 Hours Postdose (AUC0-24) of Drospirenone | Predose on Day 1 up to 144 days postdose
  PK: AUC0-24 of Drospirenone
PK: Maximum Observed Concentration (Cmax) of Drospirenone | Predose on Day 1 up to 144 days postdose
  PK: Cmax of Drospirenone
PK: Time of Maximum Observed Concentration (Tmax) of Drospirenone | Predose on Day 1 up to 144 days postdose
  PK: Tmax of Drospirenone

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Qps-Mra, Llc, South Miami, Florida
  - ICON Early Phase Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No